CLINICAL TRIAL: NCT02412904
Title: Phase 4 Study Comparing Recombinant Follicle Stimulating Hormone (rFSH) or Ultra-pure to HMG in Patients Submitted to IVF Using Gnrh Antagonist
Brief Title: Randomized Controlled Trial Comparing Embryonic Quality in rFSH Versus hMG in IVF Protocol With GnRH Antagonist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Center for Human Reproduction (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130120
Record Dates: First submitted 2013-11-05; First posted 2015-04-09 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Infertility
Keywords: follicular stimulating hormone; human menopausal gonadotrophin; Recombinant follicular stimulating hormone (rFSH); Gonadotrophin releasing hormone (GnRH) antagonists; GnRH agonist; in vitro fertilization; controled ovarian stimulation; number of mature oocytes
MeSH Terms: conditions — Infertility | interventions — follitropin beta; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- drug to ovulation induction: rFSH (Other): Patients submitted to IVF that will use rFSH (Puregon®, Organon Ltd., Ireland) for ovarian stimulation
  Interventions: Drug: rFSH
- drug to ovulation induction :HMG (Other): Patients submitted to IVF that will use hMG (Menopur®, Ferring Pharmaceuticals, Denmark) for ovarian stimulation
  Interventions: Drug: HMG

INTERVENTIONS:
Drug: rFSH — the patients will be asked to schedule an ultrasound in the first three days of the menstrual cycle and starts the ovarian stimulation with the previous randomized selected gonadotropin (rFSH or hMG) using a dose between 150 - 300 IU according with their AMH and antral follicle count (AFC). This dose will be maintained until day 6 of stimulation, when a second ultrasound will be performed and the GnRH antagonist will be initiated and continued until the end of the cycle. Seriated ultrasounds will be performed each two days
  Other Names: Puregon®, Organon Ltd., Irlanda
  Arms: drug to ovulation induction: rFSH
Drug: HMG — the patients will be asked to schedule an ultrasound in the first three days of the menstrual cycle and starts the ovarian stimulation with the previous randomized selected gonadotropin (rFSH or hMG) using a dose between 150 - 300 IU according with their AMH and AFC. This dose will be maintained until day 6 of stimulation, when a second ultrasound will be performed and the GnRH antagonist will be initiated and continued until the end of the cycle. Seriated ultrasounds will be performed each two days
  Other Names: Menopur
  Arms: drug to ovulation induction :HMG

SUMMARY:
rFSH and HMG are both used to controlled ovarian stimulation for patients submitted to IVF. However, there is a debate in the literature which one is better to induce ovulation in patients receiving GnRH antagonist to block premature Luteinizing Hormone (LH) secretion.

The investigators propose a Randomized Clinical Trial (RCT) to investigate the differences among recombinant FSH and HMG in patients submitted to IVF using GnRH antagonists.

DETAILED DESCRIPTION:
To compare embryonic quality and other clinical outcomes when using human menopause gonadotropin (hMG) or recombinant follicle stimulating hormone (rFSH) to the ovarian stimulation in IVF cycles with the GnRH antagonist protocol.

Design: open randomized single center study with infertile patients submitted to IVF comparing IVF outcomes between hMG and rFSH when controlled with GnRH antagonist.

Setting: A single private center of reproductive medicine in association with Universidade Federal do Rio Grande do Sul.

Patients: Infertile women with normal ovarian reserve with IVF indication. Intervention: The patients were randomized in two groups, 85 received rFSH and 83 received hMG to ovulation induction, both groups used GnRH antagonist to prevent ovulation.

Main Outcome Measure: Total embryonic score and best embryonic score. Secondary outcomes: Total dose of gonadotropins, number and size of follicles in the end of the stimulation, number of mature oocytes, number of embryos, pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 40 y
* infertile
* submitted to IVF
* no hormonal disease
* normal FSH (< 10)
* anti-mullerian hormone (AMH) > 1 ng and < 10 ng
* both ovaries
* only first or second IVF

Exclusion Criteria:

* thyroid-stimulating hormone (TSH), prolactin (PRL) altered
* endometrioma
* ovarian tumor or cysts
* previous Ovarian Hyperstimulation Syndrome (OHSS)
* severe male factor

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Embryo quality - score of embryo quality in the model od the Graduated Embryo Score (GES) | 3 to 5 days after the ovarian punction
  The embryo evaluation will be performed on day three after fertilization based on the Graduated Embryo Score (GES). It will be performed three evaluations occurring at 16 - 18 hours, 25 - 27 hours and 64 - 67 hours post insemination, by the same embryologist (DS) The score is composed by the following criteria: nucleolar alignment along pronuclear axis, regular cleavage and degree of fragmentation at the first cell division, and cell number and morphology on day 3 after fertilization. The score ranges from 20 to 100 per embryo.

SECONDARY OUTCOMES:
number of follicles graduated by size in groups of 13-14mm; 15-16mm and more than 17mm | 10 to 13 days after the IVF protocol starts
total number of units of gonadotrophins used to ovarian stimulation | 10 to 13 days after the IVF protocol starts
number of oocytes retrieved (MII) | 10 to 13 days after the IVF protocol starts
number of embryos | 3 to 5 days after the ovarian punction

CONTACTS AND LOCATIONS:
Overall Officials: João SL Cunha Filho, Dr, Principal Investigator — Centro de Reproduçao Humana Insemine
Locations (1):
- Centro de Reproduçao Humana Insemine, Porto Alegre, RGS, Brazil